CLINICAL TRIAL: NCT03186092
Title: Effects of Respiratory Muscle Training on Respiratory Muscle Strength, Functional Capacity and Quality of Life in Pulmonary Hypertension
Brief Title: Effects of Training in Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Profa. Dra. Vera Lúcia dos Santos Alves, PhD Health Science and Head of Cardiorespiratory Physiotherapy, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 64139317.5.0000.5479
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2019-11

CONDITIONS: Respiratory Muscle Strength
Keywords: Respiratory muscle strength; Pulmonary hypertension; Respiratory muscle training
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The equipment is the same for both groups. The change is internal, in the placebo group, patients train without a spring that imposes the load for respiratory muscle training.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): inspiratory muscle training with load
  Interventions: Other: respiratory muscle training
- Control Group (Sham Comparator): unloaded inspiratory muscle training
  Interventions: Other: sham muscle training

INTERVENTIONS:
Other: respiratory muscle training — The TMI protocol will be performed with POWERbreathe Line Plus (POWERbreathe International Ltd. Warwickshire, England) linear loader with resistance load of 30% of maximal inspiratory pressure (PImax) value for a period of 12 weeks, 7 times at Week, 30 min / day, one of the times in the week with the supervision of the researcher and, on the other six days of the week, patients will perform IMT at their homes, having as a control a records record of the protocol that will be delivered to each patient To record the time and duration of the exercise. At the end of each week, patients will be reevaluated for MIP, so that the load values are regulated according to the possible increase in inspiratory muscle strength. The data collection will be performed by a single evaluator and the patients will be properly oriented on the procedures to be performed.
  Arms: Intervention Group
Other: sham muscle training — sham comparator
  Arms: Control Group

SUMMARY:
Pulmonary hypertension (HP) is a progressive pathological condition presents with vascular changes in the lung. Cardiopulmonary changes in PH are considered the main limiting factor, however, it is known that the muscular alterations potentiate the symptomatology. Several HP factors and mechanisms have an impact on peripheral and respiratory muscle changes, so, specifically, respiratory muscles are also altered in patients with PH.

In the face of respiratory muscle weakness, inspiratory muscle training (IMT) has been shown to increase respiratory muscle strength and functional capacity in chronic conditions such as obstructive pulmonary disease (COPD) and heart failure (HF).

The objective of this study is to test whether a 12-week TMI protocol is capable of impacting functional capacity, respiratory muscle strength, spirometric values and quality of life in patients with PH.

DETAILED DESCRIPTION:
Pulmonary hypertension (HP) is a progressive pathological condition that HP presents with vascular changes in the lung that cause proliferative and obstructive remodeling promoting vasoconstriction with a consequent increase in pulmonary vascular resistance (PVR).

Cardiopulmonary changes in PH are considered the main limiting factor, however, it is known that the muscular alterations potentiate the symptomatology. Several HP factors and mechanisms have an impact on peripheral and respiratory muscle changes, such as: decreased cardiac output, hypoxemia, inflammation, increased insulin resistance, altered autonomic nervous system (ANS) response, and muscle disuse. These factors imply alteration of fiber type, atrophy, capillary vascular reduction, reduction of oxidative capacity, endothelial dysfunction and decreased muscle excitability by ANS.

Specifically, respiratory muscles are also altered in patients with PH. For the treatment of PH, in addition to optimized drug therapy, studies have demonstrated the effects of physical exercise for this population. Although there is no consensus about the best exercise modality, duration, frequency or intensity, physical training promotes benefits in exercise capacity, maximal oxygen capacity (VO2peak) and quality of life. The most recent European guideline [3] recommends supervised exercise in patients with PH who are clinically stable with optimized drug therapy (evidence grade IIa, Level B), but patients often do not have access to supervised physical rehabilitation programs, which Practice a challenge.

In the face of respiratory muscle weakness, inspiratory muscle training (IMT) has been shown to increase respiratory muscle strength and functional capacity in chronic conditions such as obstructive pulmonary disease (COPD) and heart failure (HF). At HP, the study by Saglam M et al., 2015 demonstrates improvement of respiratory muscle strength and functional capacity, resulting in decreased dyspnea and fatigue in PH patients who performed the IMT protocol during six weeks of outpatient training.

The objective of this study is to test whether a 12-week TMI protocol is capable of impacting functional capacity, respiratory muscle strength, spirometric values and quality of life in patients with PH.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary hypertension (PAP m ≥ 25mmHg and PAOP <15mmHg);
* both sexes and age greater than or equal to 18 years;
* Clinically stable with optimized and unchanged daily drug therapy in the last three months;
* agree to participate in the study by signing a free and informed consent form

Exclusion Criteria:

* Down's syndrome
* COPD
* Severe ischemic heart disease
* Left heart failure
* Cor pulmonale
* Cognitive Disorders
* Orthopedic problems that interfere with assessments and interventions
* Emergency or elective surgical intervention during the protocol
* Pulmonary infectious process during the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle strength | 3 months
  Inspiratory Muscle strength
Walk test | 3 months
  6 minute distance walk test

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Casa of Sao Paulo Medical School, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hoeper MM, Bogaard HJ, Condliffe R, Frantz R, Khanna D, Kurzyna M, Langleben D, Manes A, Satoh T, Torres F, Wilkins MR, Badesch DB. Definitions and diagnosis of pulmonary hypertension. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D42-50. doi: 10.1016/j.jacc.2013.10.032. PMID 24355641
- [Result] Simonneau G, Gatzoulis MA, Adatia I, Celermajer D, Denton C, Ghofrani A, Gomez Sanchez MA, Krishna Kumar R, Landzberg M, Machado RF, Olschewski H, Robbins IM, Souza R. Updated clinical classification of pulmonary hypertension. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D34-41. doi: 10.1016/j.jacc.2013.10.029. PMID 24355639
- [Result] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Respir J. 2015 Oct;46(4):903-75. doi: 10.1183/13993003.01032-2015. Epub 2015 Aug 29. PMID 26318161
- [Result] Ehlken N, Verduyn C, Tiede H, Staehler G, Karger G, Nechwatal R, Opitz CF, Klose H, Wilkens H, Rosenkranz S, Halank M, Grunig E. Economic evaluation of exercise training in patients with pulmonary hypertension. Lung. 2014 Jun;192(3):359-66. doi: 10.1007/s00408-014-9558-9. Epub 2014 Mar 8. PMID 24609926
- [Result] Gosselink R, De Vos J, van den Heuvel SP, Segers J, Decramer M, Kwakkel G. Impact of inspiratory muscle training in patients with COPD: what is the evidence? Eur Respir J. 2011 Feb;37(2):416-25. doi: 10.1183/09031936.00031810. PMID 21282809
- [Result] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Result] Neder JA, Andreoni S, Lerario MC, Nery LE. Reference values for lung function tests. II. Maximal respiratory pressures and voluntary ventilation. Braz J Med Biol Res. 1999 Jun;32(6):719-27. doi: 10.1590/s0100-879x1999000600007. PMID 10412550
- [Result] Simonneau G, Galie N, Rubin LJ, Langleben D, Seeger W, Domenighetti G, Gibbs S, Lebrec D, Speich R, Beghetti M, Rich S, Fishman A. Clinical classification of pulmonary hypertension. J Am Coll Cardiol. 2004 Jun 16;43(12 Suppl S):5S-12S. doi: 10.1016/j.jacc.2004.02.037. PMID 15194173
- [Result] Mereles D, Ehlken N, Kreuscher S, Ghofrani S, Hoeper MM, Halank M, Meyer FJ, Karger G, Buss J, Juenger J, Holzapfel N, Opitz C, Winkler J, Herth FF, Wilkens H, Katus HA, Olschewski H, Grunig E. Exercise and respiratory training improve exercise capacity and quality of life in patients with severe chronic pulmonary hypertension. Circulation. 2006 Oct 3;114(14):1482-9. doi: 10.1161/CIRCULATIONAHA.106.618397. Epub 2006 Sep 18. PMID 16982941
- [Result] Saglam M, Arikan H, Vardar-Yagli N, Calik-Kutukcu E, Inal-Ince D, Savci S, Akdogan A, Yokusoglu M, Kaya EB, Tokgozoglu L. Inspiratory muscle training in pulmonary arterial hypertension. J Cardiopulm Rehabil Prev. 2015 May-Jun;35(3):198-206. doi: 10.1097/HCR.0000000000000117. PMID 25909652